CLINICAL TRIAL: NCT06037707
Title: Incidence of Thromboembolism in COVID-19 Infection in the ICU: a Retrospective Cohort Analysis
Brief Title: Thromboembolic Complications in COVID-19 Patients in Intensive Care Unit
Acronym: COVID-19TC
Status: Completed | Type: Observational
Sponsor: Ayse Zeynep Turan (Other)
Responsible Party: Sponsor-Investigator, Ayse Zeynep Turan, Principle Investigator, Derince Training and Research Hospital
Organization: Derince Training and Research Hospital (Other)
Other Study IDs: DerinceTRH-07
Record Dates: First submitted 2023-09-01; First posted 2023-09-14 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: COVID-19-Associated Thromboembolism
Keywords: COVID-19; thromboembolism; Variants of COVID-19
MeSH Terms: conditions — COVID-19; Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Ancestral variant: Ancestral variant is the first subtype of SARS CoV-2 virus which is the agent of first COVID-19 infection in Wuhan. Thromboembolic complications of this group were detected among patients which were infected with ancestral variant of COVID-19
- Delta Variant: Delta variant is the subtype of SARS CoV-2 virus which is first COVID-19 subtype identified in India. Thromboembolic complications of this group were detected among patients which were infected with delta variant of COVID-19
- Alpha variant: Alpha variant is the subtype of SARS CoV-2 virus which is first identified COVID-19 subtype in United Kingdom. Thromboembolic complications of this group were detected among patients which were infected with alpha variant of COVID-19
- Other variants: Other variants is the subtype of SARS CoV-2 virus which were identified in Brazil, South Africa..etc. Thromboembolic complications of this group were detected among patients which were infected with alpha variant of COVID-19

SUMMARY:
The present study aims to determine frequency of thromboembolic complications and the underlying causes of this complication of the patients who admitted to the intensive care unit diagnosed with COVID-19.

DETAILED DESCRIPTION:
Patients diagnosed with COVID-19 infection and admitted to the ICU were recruited. Demographic information, comorbidities, length of ICU stay, some laboratory data,thromboembolic complications of the patients were recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were infected with COVID-19 and admitted to the intensive care unit between the time of March 2020-December 2021

Exclusion Criteria:

* who is under 18 years old.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study Population of the present study is all of the patients diagnosed with COVID-19 and admitted to the intensive care units at Derince Training and Research Hospital at the time of between 1-March-2020 and 31-December-2021in
Sampling Method: Probability Sample
Enrollment: 484 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Rate of thromboembolic complications among patients who effected from different variants of COVID-19 Disease | During the entire intensive care stay up to 1 day
  Both arterial and venous thromboembolic events were detected

SECONDARY OUTCOMES:
Rate of thromboembolic complications of COVID-19 disease in critically ill patients | During the entire intensive care stay up to 1 day
  Both arterial and venous thromboembolic events were detected
Rate of thromboembolic complications according to anticoagulant therapy | During the entire intensive care stay up to 1 day
  Antithrombotic therapy of each patient was recorded
What is the rate of thromboembolism according to the comorbidities | During the entire intensive care stay up to 1 day
  Comorbidities of each patient were recorded from the patients records.

CONTACTS AND LOCATIONS:
Overall Officials: Berna Karakoyun Lacin, Prof., Principal Investigator — Health and Science University Hamidiye Institute of Health Sciences
Locations (1):
- Derince Research and Training Hospital, Kocaeli, Derince, Turkey (Türkiye)